CLINICAL TRIAL: NCT01385709
Title: The Influence of the Menstrual Cycle on Lithium and Sertraline Blood Levels
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 0310006393
Record Dates: First submitted 2011-06-13; First posted 2011-06-30 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Bipolar Affective Disorders; Cyclothymic Disorder; Schizoaffective Disorder; Major Depressive Disorder; Dysthymic Disorder; Obsessive-Compulsive Disorder; Panic Disorder; Posttraumatic Stress Disorder; Premenstrual Dysphoric Disorder; Social Anxiety Disorder
Keywords: Lithium; Sertraline
MeSH Terms: conditions — Cyclothymic Disorder; Psychotic Disorders; Depressive Disorder, Major; Dysthymic Disorder; Obsessive-Compulsive Disorder; Panic Disorder; Stress Disorders, Post-Traumatic; Premenstrual Dysphoric Disorder; Phobia, Social

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood will be drawn.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sertraline: Therefore, patients who are already taking psychotropic medications, and therefore are currently in treatment for a psychiatric illness, will be recruited. The specific psychiatric diagnoses anticipated in the subject pool include the conditions that sertraline is indicated to treat, including Bipolar Affective Disorders, Cyclothymic Disorder, Schizoaffective Disorder, Major Depressive Disorder, Dysthymic Disorder, Obsessive-Compulsive Disorder, Panic Disorder, Posttraumatic Stress Disorder, Premenstrual Dysphoric Disorder, and Social Anxiety Disorder. Patients must be female, between the ages of 18-40, taking either sertraline on a daily basis for at least one week. Exclusion criteria include 1) currently pregnant or breastfeeding, 2) concurrent use of any form of hormonal birth control, including oral contraceptive pills, Norplant or Depo-provera, 3) hepatic or renal disease, 4) irregular menstrual cycles.
- Lithium: Therefore, patients who are already taking psychotropic medications, and therefore are currently in treatment for a psychiatric illness, will be recruited. The specific psychiatric diagnoses anticipated in the subject pool include the conditions that lithium is indicated to treat, including Bipolar Affective Disorders, Cyclothymic Disorder, Schizoaffective Disorder, Major Depressive Disorder, Dysthymic Disorder, Obsessive-Compulsive Disorder, Panic Disorder, Posttraumatic Stress Disorder, Premenstrual Dysphoric Disorder, and Social Anxiety Disorder. Patients must be female, between the ages of 18-40, taking lithium on a daily basis for at least one week. Exclusion criteria include 1) currently pregnant or breastfeeding, 2) concurrent use of any form of hormonal birth control, including oral contraceptive pills, Norplant or Depo-provera, 3) hepatic or renal disease, 4) irregular menstrual cycles.

SUMMARY:
The aim of this study is to determine whether blood levels of lithium or sertraline are affected by different phases of the menstrual cycle and whether there is an effect on psychiatric symptoms. Subjects are seen for two visits: one visit during the luteal phase and one visit during the follicular phase of the menstrual cycle. On each visit, they will fill out a depression, anxiety and mania rating scale. Also at each visit a 20mL blood sample will be drawn to measure progesterone level and either a lithium or sertraline level, depending on which medication the patient takes. The primary hypothesis in this study is that blood levels of lithium and sertraline will be significantly lower in women during the luteal phase of the menstrual cycle than during the follicular phase. Examination will also be made of whether symptoms will increase in severity during the luteal phase as compared to the follicular phase. The investigators expect a negative linear association between symptom severity and blood level, i.e. expect symptom severity to worsen as blood levels of lithium or sertraline decrease.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 year old female
* women currently taking Lithium or Sertraline

Exclusion Criteria:

* currently pregnant or breastfeeding
* concurrent use of any form of hormonal birth control, including oral contraceptive pills, Norplant or Depo-provera
* hepatic or renal disease
* irregular menstrual cycles.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The specific psychiatric diagnoses anticipated in the subject pool include the conditions that lithium and sertraline are indicated to treat, including Bipolar Affective Disorders, Cyclothymic Disorder, Schizoaffective Disorder, Major Depressive Disorder, Dysthymic Disorder, Obsessive-Compulsive Disorder, Panic Disorder, Posttraumatic Stress Disorder, Premenstrual Dysphoric Disorder, and Social Anxiety Disorder.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2008-08; Primary Completion 2012-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
blood levels of lithium or sertraline | 5-9 days after menstrual cycle onset
  Determine whether the blood levels of lithium or sertraline are affected by different phases of the menstrual cycle.
Fluctuations in symptom severity | 5-9 days after onset of menstrual cycle
  Determine whether there is a fluctuation in symptom severity during different phases of the menstrual cycle.
blood levels of lithium or sertraline | 5-9 days before onset of next menstrual cycle
  Determine whether the blood levels of lithium or sertraline are affected by different phases of the menstrual cycle.
Fluctuations in symptom severity | 5-9 days before onset of next menstrual cycle
  Determine whether there is a fluctuation in symptom severity during different phases of the menstrual cycle.

SECONDARY OUTCOMES:
Correlations between Symptom Severity and Blood Levels of Drugs | 5-9 days after onset of menstrual cycle
  Determine whether there is a correlation between blood levels of lithium or sertraline and symptom severity during different phases of the menstrual cycle.
Correlations between Symptom Severity and Blood Levels of Drugs | 5-9 days before onset of next menstrual cycle
  Determine whether there is a correlation between blood levels of lithium or sertraline and symptom severity during different phases of the menstrual cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Mallay B Occhiogrosso, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- See also: Weill Cornell Medical College website — http://med.cornell.edu